CLINICAL TRIAL: NCT01118871
Title: A Randomised, Open Label, Prospective Study to Assess Two Different Therapeutic Strategies Following First Treatment Failure in HIV-1 Infected Subjects
Brief Title: The First Failure Study
Acronym: FAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAST1.0
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2010-07

CONDITIONS: HIV; HIV Infections
Keywords: Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Drug: Darunavir, Ritonavir, Truvada
- NRTI sparing arm (Experimental)
  Interventions: Drug: Darunavir, Ritonavir and Etravirine

INTERVENTIONS:
Drug: Darunavir, Ritonavir, Truvada — Darunavir 800 mg daily Ritonavir 100 mg daily Tenofovir 245 mg daily Emtricitabine 200 mg daily
  Other Names: Prezista; Norvir; Truvada
  Arms: Standard of care
Drug: Darunavir, Ritonavir and Etravirine — Darunavir 800 mg daily Ritonavir 100 mg daily Etravirine 400 mg once daily
  Other Names: Prezista; Norvir; Intelence
  Arms: NRTI sparing arm

SUMMARY:
The purpose of this study is to look at two different antiretroviral treatment options in individuals who are about to commence their second antiretroviral treatment.

This study will assess important clinical and laboratory differences between these two therapeutic options. Potential differences include: differences in body fat distribution, in lipid parameters, in adherence and in neurocognitive (brain) function. This study is looking to show differences in body fat distribution between the two study treatment arms. Differences in lipids, viral load, adherence, cardiac and bone biomarkers and neurocognitive function will also be assessed. There is also a lumbar puncture sub study participants can also take part in.

The total duration of involvement in the trial will be up to 96 weeks (approximately 2 years) plus a screening visit 1 - 4 weeks prior to the start of the study. Including visit the clinic on 12 occasions (screening visit, baseline visit, weeks 2, 4, 8, 12, 24, 36, 48, 64, 80 and 96)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* over 18 years of age
* signed informed consent
* currently receiving a stable antiretroviral regimen comprising of:
* two or more licensed NRTIs
* one licensed NNRTI or boosted protease inhibitor
* no previous protease inhibitor resistance documented on HIV-1 genotypic resistance testing
* failure of current antiretroviral regimen due to:
* toxicity, intolerance or virological failure if receiving an NNRTI containing regimen at screening
* toxicity or intolerance if receiving a boosted-protease inhibitor regimen at screening (with plasma HIV RNA < 400 copies/mL at screening)
* willing to modify antiretroviral therapy, in accordance with the randomisation assignment
* no previous exposure to etravirine
* subjects in good health upon medical history, physical exam, and laboratory testing in the opinion of the investigator
* have no serologic evidence of active HBV infection evidenced by negative hepatitis B surface antigen
* female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must practice contraception as follows from screening through completion of the study:
* barrier contraceptives (condom, diaphragm with spermicide)
* IUD or Depo PLUS a barrier contraceptive
* female subjects of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

* current alcohol abuse or drug dependence
* pregnancy
* active opportunistic infection or significant co-morbidities
* current prohibited concomitant medication
* a likelihood of diminished response to any of the study treatment arms, in the opinion of the investigator, based on HIV genotypic resistance testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in peripheral and central adipose tissue | week 48 and 96
  As measured by DEXA, between treatment arms.

SECONDARY OUTCOMES:
Percentage of patients <50 copies HIV-1 RNA/mL | 96 weeks
  At all study points to weeks 48 and 96 between treatment arms.
Mean change from baseline of absolute CD4+ T cell count | 96 weeks
  between treatment arms
Time to change in randomly assigned therapy | 96 weeks
  between treatment arms
Mean change from baseline Lipodystrophy Case Definition score | 96 weeks
  Between treatment arms
Mean change from baseline in fasting lipid and glycaemia parameters | 96 weeks
  between treatment arms
Mean change from baseline in cardiac and bone biomarker levels | Week 96
  between treatment arms
• Comparison of total number of patients with any serious adverse events (SAEs), and the cumulative incidence of SAEs | 96 week s
  Between the treatment arms
Patterns of genotypic HIV resistance associated with virological treatment failure | 96 weeks
  Across the treatment arms
Describe aspects of immune reconstitution disease (IRD) | 96 weeks
  Across the treatment arms
Comparison of quality of life and results of adherence questionnaires | 96 weeks
  Between the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MB ChB, Principal Investigator — Imperial College London
Locations (1):
- St. Mary's Hospital, London, United Kingdom